CLINICAL TRIAL: NCT06215404
Title: Effects of Different Fluid Management Strategies on Blood Loss, Inflammatory Response, and Major Organ Sequelae in Liver Transplantation
Brief Title: Fluid Management Strategies on Blood Loss in Liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202308015MINC
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Liver Transplant
Keywords: fluid management; blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal group (Active Comparator): stroke volume variation < 10%
  Interventions: Other: Liberal group
- restrictive group (Experimental): stroke volume variation < 18%
  Interventions: Other: restrictive group

INTERVENTIONS:
Other: Liberal group — Fluid challage to keep stroke volume variation < 10%
  Arms: Liberal group
Other: restrictive group — Fluid challage to keep stroke volume variation < 18%
  Arms: restrictive group

SUMMARY:
During liver transplantation, due to the complexity of the operation and abnormal coagulation function, there may be a large amount of bleeding and corresponding blood transfusion. Excessive blood transfusion will increase pulmonary complications and affect the prognosis. Infusion management to reduce bleeding is a very important issue in liver transplant surgery. Restrictive infusion management can effectively reduce the amount of bleeding in liver transplantation, but it remains unclear whether it will cause sequelae in other major organs.

The investigators plan to study different infusion goals and strategies in liver transplant surgery using a randomized group model, using the PiCCO (Pulse Contour Cardiac Output) cardiopulmonary volume monitor, and setting the stroke volume variation (SVV) as the macroscopic circulation.The purpose of this study was to divide it into restrictive and liberal groups to explore the impact on liver transplantation bleeding volume and inflammatory response as well as postoperative lung and renal function, and to collect statistics on clinical care and postoperative sequelae (pulmonary liver, renal function impairment, etc.) in order to develop the most appropriate infusion management strategy in liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* end stage liver disease
* age between 18y/o to 75 y/o
* expected to recieve to receive liver transplantation

Exclusion Criteria:

* arrythmia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
blood loss intraoperatively | during the operation
  blood loss intraoperatively in liver transplant

SECONDARY OUTCOMES:
Lung injury biomarker | from biginning of the operation to postoprative day 1
  serum Clara Cell Protein (CC16)
Kidney injury biomarker | from biginning of the operation to postoprative day 1
  serum Neutrophil Gelatinase Associated Lipocalins (NGALs)
Influammatory reponses | from biginning of the operation to postoprative day 1
  IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Cheng Chan, M.D.,PhD., Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No